CLINICAL TRIAL: NCT02548143
Title: Phase 3 Study of Safety and Efficacy of Coagulation Factor VIIa (Recombinant) for Prevention of Excessive Bleeding in Congenital Hemophilia A/B Patients With Inhibitors to Factor VIII/IX Undergoing Elective Surgery/Other Invasive Procedures
Brief Title: LR769 in Congenital Hemophilia Patients With Inhibitors Undergoing Elective Surgery or Invasive Procedures
Acronym: PerSept3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Collaborators: LFB USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LFB-FVIIa-008-14
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coagulation Factor VIIa (Recombinant) (Experimental): A dose of 75 μg/kg (minor surgery or invasive procedure) or 200 μg/kg (major surgery or major invasive procedure) of LR769 will be administered as an initial intravenous (IV) bolus dose of LR769 within ≤2 minutes before the surgical incision or start of the invasive procedure. For both minor and major procedures, the initial dose will be followed by repeated administration of 75 µg/kg of LR769 every 2 hours (±5 minutes) for the first 48 hours after completion of the procedure and then as per the dosing schedules in the protocol for major or minor surgeries or invasive procedures. The minimum duration of LR769 treatment for major procedures will be 5 days, and for minor procedures 2 days except for certain procedures that may not require this duration of treatment.
  Interventions: Biological: Coagulation Factor VIIa (Recombinant)

INTERVENTIONS:
Biological: Coagulation Factor VIIa (Recombinant) — LR769

SUMMARY:
The purpose of this study, PerSept 3, is to evaluate LR769 for the prevention of excessive bleeding and achievement of hemostasis in congenital hemophilia A or B patients who have inhibitors to Factor VIII or Factor IX , are aged 6 months to 75 years, inclusive; and who are undergoing elective surgical or other invasive procedures. Administration of LR769 will be performed just prior to surgery/procedure and will be repeated during and after the surgery/procedure to achieve and maintain adequate hemostasis as determined by the investigator's judgment.

DETAILED DESCRIPTION:
This study is an international, multicenter, single-arm, Phase 3 study. Patients aged 6 months to 75 years, inclusive, who have congenital hemophilia A or B with inhibitors to Factor VIII or Factor IX and who are scheduled for an elective surgical or other invasive procedure will be enrolled. Both major and minor surgical or other invasive procedures are allowed in the study.

Initial Treatment: Regardless of procedure, patients who meet all eligibility criteria will receive an initial intravenous (IV) bolus dose of LR769 within ≤2 minutes before the surgical incision or start of the invasive procedure. For a minor elective surgery or other minor invasive procedure, a dose of 75 μg/kg will be used as the initial dose; for a major elective surgery or other major invasive procedure, a dose of 200 μg/kg of LR769 will be used as the initial dose. For both minor and major procedures, administration will be repeated no more frequently than every 2 hours (±5 minutes) at a dose of 75 μg/kg during and after surgery or invasive procedure.

Treatment for Major Surgical Procedures: The initial dose of LR769 will be followed by repeated administration of 75 µg/kg of LR769 every 2 hours (±5 minutes) for the first 48 hours after completion of the procedure. The minimum duration of LR769 treatment for major procedures will be 5 days and dosing frequency will be followed according to the guidelines specified in the protocol.

Treatment for Minor Surgical or Other Invasive Procedures: The initial dose of LR769 will be followed by repeated administration of 75 µg/kg of LR769 every 2 hours (±5 minutes) for the first 48 hours. The minimum duration of LR769 infusion for minor procedures will be 2 days, except for certain procedures that may not require this duration of treatment to achieve hemostasis as noted in the protocol. Dosing frequency will be according to the guidelines specified in protocol for minor surgical or other invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study:

1. be male with a diagnosis of congenital hemophilia A or B of any severity
2. have one of the following:

   1. a positive inhibitor test Bethesda Unit (BU) ≥5 (as confirmed at screening by the institutional lab), OR
   2. a BU <5 but expected to have a high anamnestic response to FVIII or FIX, as demonstrated from the patient's medical history, precluding the use of FVIII or FIX products to treat or prevent bleeding, OR
   3. a BU <5 but expected to be refractory to increased dosing of FVIII or FIX, as demonstrated from the patient's medical history, precluding the use of FVIII or FIX products to treat or prevent bleeding episodes
3. be ≥6 months to ≤75 years of age; different age restrictions may apply per local regulation and ethical considerations (enrollment of children <12 years of age will not begin until after review of data from the PERSEPT 2 study by the DMC)
4. be scheduled for an elective surgical or other invasive procedure
5. be capable of understanding and willing to comply with the conditions of the protocol OR in the case of a patient <18 years of age, parent(s)/legal guardian(s) must be capable of understanding and willing to comply with the conditions of the protocol
6. have read, understood, and provided written Informed Consent (patient and/or parent(s)/legal guardian(s) if the patient is <18 years of age) or Assent, if applicable

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. have any coagulation disorder other than hemophilia A or B
2. be immunosuppressed (ie, the patient should not be receiving systemic immunosuppressive medication; cluster of differentiation 4 (CD4) counts at screening should be >200/µL)
3. known intolerance to LR769 or any of its excipients
4. currently receiving immune tolerance induction (ITI) therapy
5. have a known allergy or hypersensitivity to rabbits
6. have a platelet count<100,000/µL
7. have received an investigational drug within 30 days of the planned first LR769 administration , or is expected to receive such drug during participation in this study (with the exception of patients who are or were participating in another LR769 study, eg, a study assessing the treatment of bleeding episodes with LR769)
8. have a clinically relevant hepatic (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN)) and/or renal impairment (creatinine >2 times the ULN)
9. have a history of arterial and/or venous thromboembolic events (such as myocardial infarction, ischemic strokes, transient ischemic attacks, deep venous thrombosis (DVT) or pulmonary embolism (PE)) within 2 years prior to the planned first dose of LR769, uncontrolled arrhythmia, or current New York Heart Association (NYHA) functional classification score of stages II - IV
10. have an active malignancy (those with non-melanoma skin cancer are allowed)
11. have any life-threatening disease or other disease or condition which, according to the investigator's judgment, could imply a potential hazard to the patient, or interfere with the trial participation or trial outcome (eg, a history of non-responsiveness to bypassing products)
12. be using aspirin, NSAIDS, herbs, natural medications, or other drugs with platelet inhibitory properties within one week prior to surgery and for the duration of treatment with LR769
13. have active gastric or duodenal ulcer disease

Ages: 6 Months to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2017-08-06 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Escobar, MD, Principal Investigator — Memorial Hermann Texas Medical Center
Locations (9):
- UT Southwestern Medical Center, Dallas, Texas, United States
- Dr. Jose Eleuterio Gonzalez Monterrey University Hospital, Monterrey, Nuevo León, Mexico
- Hematology Research Center of the Russian Academy of Medical Sciences, Moscow, Russia
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Hemophilia Comprehensive Care, Parktown, Gauteng
  - Worthwhile Clinical Trials, Lakeview Hospital, Benoni
- University and Polytechnic Hospital La Fe, Hemostasis and Thrombosis Unit, Valencia, Spain
- Ukraine (3):
  - City Scientific-Practical center for diagnosics, Kiev
  - National Specialized Children's Hospital OKHMATDYT, Centre for Hemostatic Pathology, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine, Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg): Major surgical procedures were those that usually required ≥5 days of factor replacement in hemophilia patients with inhibitors and typically involved entry into a body cavity and/or organ removal or similarly complex procedures.
  A dose of 200 μg/kg of LR769 administered within ≤2 minutes of the onset of the procedure was used as the initial dose before the surgical incision or start of the invasive procedure. The initial dose was followed by repeated administration of 75 μg/kg of LR769 every 2 hours (±5 minutes) for the first 48 hours after completion of the procedure. After 48 hours, dosing continued at 75 μg/kg of LR769 (not more frequently than every 2 hours) as follows:
  Days 3-4: Intervals up to every 4 hours; Days 5-6: intervals up to every 6 hours; Days 7-10: Intervals up to every 8 hours; Days 11 to last administration of LR769: Intervals up to every 12 hours.
- Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg): Minor surgical or other invasive procedures were those that usually required <5 days of factor replacement and usually involved the skin, mucous membranes, or superficial connective tissue. The minimum duration of LR769 infusion for minor procedures was 2 days. For less invasive procedures, the patient may have been treated for ≤48 hours if the investigator/designee determined a shorter duration was sufficient to achieve hemostasis.
  A dose of 75 μg/kg of LR769 administered within ≤2 minutes of the onset of the procedure was used as the initial dose before the surgical incision or start of the invasive procedure. The initial dose was followed by repeated administration of 75 μg/kg of LR769 every 2 hours (±5 minutes) for the first 48 hours. From Day 3, dosing could continue at 75 μg/kg of LR769 at intervals of up to every 24 hours, but not more frequently than every 2 hours.
Period: Overall Study
Arm/Group | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg)
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (20.19) | 16.0 (15.52) | 25.0 (19.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ukraine | 3 | 3 | 6
  South Africa | 1 | 3 | 4
  Mexico | 1 | 0 | 1
  Russia | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 54.17 (25.974) | 36.72 (21.506) | 45.44 (24.494)
Height [Mean (Standard Deviation); unit: cm] | 156.3 (22.50) | 137.8 (34.02) | 147.1 (29.13)
BMI [Mean (Standard Deviation); unit: kg/ m^2] | 20.88 (6.203) | 17.61 (2.823) | 19.24 (4.902)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Surgical or Other Invasive Procedures Defined as "Good" or "Excellent" Response to LR769 Treatment as Assessed by the Investigator, Based on the Totality of the Assessments Performed on the Patient
Description: The final assessment was performed by the investigator at the study center 48 hours after the last dose of LR769 and was based upon the totality of the assessments performed on the patient at each time point. Excellent: postoperative blood loss similar to or less than expected following this type of procedure in a patient who does not have a bleeding disorder and who is undergoing the same surgical or other invasive procedure; no blood component transfusion is required. Good: postoperative blood loss greater, but not substantially greater than expected, following this type of procedure in a patient who does not have a bleeding disorder and who is undergoing the same surgical or other invasive procedure, not explained by a surgical/medical issue other than hemophilia; no unexpected need for blood component transfusion.
Time Frame: 48 (±4) hours after the last administration of LR769
Population: Efficacy Population: All patients who received LR769 treatment, underwent a surgical or invasive procedure, and had at least one efficacy assessment.
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Arm/Group | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg)
Number analyzed (Participants) | 6 | 5
Number analyzed (Surgeries) | 6 | 5
Surgeries
  Successes | 4 | 5
  Failures | 2 | 0

2. Secondary Outcome: Percentages of Success as Defined as the Combination of "Good" and "Excellent" Responses by the Investigator or Designee
Description: Good: postoperative blood loss greater than expected following this type of procedure in a patient who does not have a bleeding disorder and who is undergoing the same surgical or other invasive procedure, not explained by a surgical/medical issue other than hemophilia; no unexpected need for blood component transfusion Excellent: postoperative blood loss similar to or less than expected following this type of procedure in a patient who does not have a bleeding disorder and who is undergoing the same surgical or other invasive procedure; no blood component transfusion is required
Time Frame: 24 hours after procedure completion
Population: as for outcome 1
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Arm/Group | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg)
Number analyzed (Participants) | 4 | 6
Number analyzed (Surgeries) | 4 | 6
Surgeries
  Successes | 4 | 6
  Failures | 0 | 0

3. Secondary Outcome: Percentages of Success as Defined as the Combination of "Good" and "Excellent" Responses by the Investigator or Designee
Description: as for outcome 2
Time Frame: 72 hours after procedure completion
Population: as for outcome 1
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Arm/Group | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg)
Number analyzed (Participants) | 5 | 2
Number analyzed (Surgeries) | 5 | 2
Surgeries
  Successes | 5 | 2
  Failures | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the time of signing of the informed consent/assent until resolution or 30 days after the last dose of LR769 or early termination, whichever came first.
Description: An AE was defined as any undesirable physical, psychological, or behavioral effect experienced by a patient or subject during participation in an investigational study, in conjunction with the use of a drug or biologic, whether or not product-related.
  Changes in coagulation parameters expected in hemophilia patients were not regarded as AEs, unless they led to clinical measures to prevent or treat any untoward events associated with the deviation of the parameter.
Arm/Group | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg)
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) (N=6) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg) (N=6)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Surgery (LR769 Initial Dose 200 μg/kg; Then 75 μg/kg) (N=6) | Minor Surgery (LR769 Initial Dose 75 μg/kg; Then 75 μg/kg) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 5 (7) | 0 (0)
Wound Secretion (Injury, poisoning and procedural complications) | 1 (2) | 2 (4)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT02548143/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02548143/SAP_001.pdf